CLINICAL TRIAL: NCT04554381
Title: Assesment of JL1 Expression in B-cell Acute Lymphoblastic Leukemia
Brief Title: Assesment of JL1 Expression in Acute Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zeinab Galal Eldeen Abdelhamid, Principal Investigator, Assiut University
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: JL1 in Acute Leukemia
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — JL1 antigen

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JL1 (Experimental): JL1 on acute leukemia
  Interventions: Biological: JL1 antigen
- JL1 and acute leukemia (Experimental): Assesment of JL1 expression on acute leukemia
  Interventions: Biological: JL1 antigen

INTERVENTIONS:
Biological: JL1 antigen — we hypothesis that JL1 can be used as an adjunctive marker for the initial diagnosis and the follow up of Acute Lymphoblastic Leukemia.

SUMMARY:
The aim of this study is to assess JL1 expression by flow cytometric immunophenotyping in patients with B-cell Acute Lymphoblastic Leukemia (ALL) and to correlate it with clinical, morphological, immunophenotypic, cytogenetic data and response to treatment.

DETAILED DESCRIPTION:
Acute Lymphoblastic Leukemia (ALL) is characterized by a rapidly progressive disease. It accounts for approximately 75% of all cases of childhood leukemias, that produces large and immature cells (20% or more lymphoblasts in the bone marrow (BM) and/or the blood) that can't carry out their normal BM function (Terwilliger and Abdul-Hay, 2017).

The main cause of ALL lies in the genetic or acquired injury to DNA of a single cell in the BM with the presence of risk factors such as radiation, benzene exposure, Down syndrome and past treatment with chemotherapeutic agents which leads to uncontrolled and exaggerated growth and accumulation of lymphoblasts which fail to function as normal blood cells. This results in blocking the production of normal blood cells and leads to anemia, thrombocytopenia and neutropenia. The most frequent signs are lymphadenopathies, hepatosplenomegaly, fever, anemia, signs of hemorrhage, and bone tenderness.

The prognostic factors of ALL include patients' factors such as age, white blood cell (WBC) count and genetic factors such as chromosome and gene changes along with the immunophenotypic characteristics of the leukemic blast cells and the individual response to therapy.

JL1 is a CD43 epitope and mucin family cell surface glycoprotein that is expressed on leukemic cells. It is expressed on hematopoietic cells at different stages of differentiation including early stage lymphoid precursors and late stage of myeloid cells. Expression patterns of JL1 antigen occurs on cell surface of leukemic cells, BM cells and phytohemagglutinin (PHA)-activated lymphocytes. Most leukemic cells usually express JL1 even in weak positive cases.

JL1 is usually expressed in about 60% of acute leukemia regardless of the lineage. It was also detected on CD34+ CD10+ lymphoid precursors and some immature myeloid cells in BM. An anti-JL1 (a monoclonal antibody that is selectively reactive with antigen in spite of the differences in the molecular weight) is mixed with a toxic substance that target the leukemic cells which leads to the emergence of its role as a therapeutic agent.

Therefore, the invistigators aim to study JL1 expression on leukemic cells in ALL patients in South Egypt Cancer Institute, as we hypothesis that it can be used as an adjunctive marker for the initial diagnosis and the follow up of ALL.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed B-cell ALL.
2. Age group: both pediatric patients (< 18 years old) and adult patients (> 18 years old) will be included in our study.

Exclusion Criteria:

1. Patients with other types of hematologic neoplasms. 2 .Relapsed patients.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-13 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation and assessment of JL1 expression in B-cell Acute Lymphoblastic Leukemia. | Baseline
  Correlatin of this marker with clinical, morphological, immunophenotypic, cytogenetic data and response to treatment.

REFERENCES:
- [Background] Terwilliger T, Abdul-Hay M. Acute lymphoblastic leukemia: a comprehensive review and 2017 update. Blood Cancer J. 2017 Jun 30;7(6):e577. doi: 10.1038/bcj.2017.53. PMID 28665419
- [Background] Park YS, Park SH, Park SJ, Kim Y, Jang KT, Ko YH, Lee MW, Huh JR, Park CS. Expression of JL1 is an effective adjunctive marker of leukemia cutis. Arch Pathol Lab Med. 2010 Jan;134(1):95-102. doi: 10.5858/2008-0699-OAR.1. PMID 20073611